CLINICAL TRIAL: NCT06628323
Title: The Neuro-VR Study: A Pilot Study Investigating an Innovative Virtual Reality-based Intervention Employing Biofeedback to Increase Tolerability and Therapy Efficacy in Psychosis
Brief Title: Neuro-VR: Augmenting a Virtual Reality-based Therapy With Biofeedback for Auditory Hallucinations
Acronym: Neuro-VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Sara Breivik Soleim, Psychologist / Research Assistant, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24010871
Record Dates: First submitted 2024-08-19; First posted 2024-10-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Auditory Hallucinations; Schizophrenia
Keywords: Virtual Reality-based therapy; Schizophrenia; Auditory Hallucinations; Neurofeedback; EEG
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality based therapy added real-time EEG-based neurofeedback (VR-NF) (Experimental): Participants in the experimental group undergo 8 sessions of a manualized virtual reality-based intervention added real-time EEG neurofeedback aiming to enhance the control and sense of power in relation to the dominant hallucinated voice. Together with the therapist, the participants create a digital representation (avatar) in virtual reality corresponding to the visual perception and sound of the voice. During therapy, the participants will be encouraged to engage in a dialogue with the avatar. While immersed in virtual reality, EEG recordings will be conducted by electrodes connected to a cap on the participants' head. Processed EEG-data will provide real-time information on the participants' brain activity associated with the emotional distress when confronted with the avatar and will be visible both to the participant and therapist. The feedback will be used to continuously adjust the intervention to the brain activity and aims to help the participant practice emotion regulation.
  Interventions: Behavioral: Virtual Reality-based Intervention employing Neurofeedback
- Virtual Reality - based therapy (Active Comparator): Participants in the control group will be offered 8 sessions of a manualized virtual reality - based therapy that follows the same principles as described in the experimental arm. Together with the therapist, the participants create a digital representation (avatar) in virtual reality that corresponds to their visual perception of and sounds like their hallucinated voice. Thoughout the therapy sessions, the participants will be encouraged to engage in a dialogue with the 'avatar', voiced by the therapist who will alternate between talking as the 'avatar' and as a supportive therapist. The therapy aims at enhancing the participants' control and feeling of power in relation to the dominant hallucinated voice. Furthermore, the therapy focuses on regulating the emotional distress associated with the hallucinated voice.
  Interventions: Behavioral: Virtual Reality-based Intervention

INTERVENTIONS:
Behavioral: Virtual Reality-based Intervention employing Neurofeedback — Virtual Reality-based intervention augmented with real-time EEG-based neurofeedback targeting auditory hallucinations in schizophrenia
  Arms: Virtual Reality based therapy added real-time EEG-based neurofeedback (VR-NF)
Behavioral: Virtual Reality-based Intervention — Virtual Reality-based intervention targeting auditory hallucinations in schizophrenia
  Arms: Virtual Reality - based therapy

SUMMARY:
The primary goal of this pilot study is to examine the feasibility and acceptability of augmenting a Virtual Reality-based intervention for treating auditory hallucinations in schizophrenia with electroencephalogram (EEG)-based neurofeedback.

The main questions it aims to answer are:

1. Is Virtual Reality -based therapy supplemented with EEG-based neurofeedback (VR-NF) a feasible and acceptable treatment for auditory hallucinations?
2. Will VR-NF show indications of being more effective than Virtual Reality-based therapy alone in reducing the severity of auditory hallucinations, improving daily functioning, and enhancing quality of life?

Researchers will compare VR-NF to Virtual Reality-based therapy alone to evaluate therapy effectiveness.

Participants will be allocated to receive 8 sessions of either VR-NF or Virtual Reality-based therapy alone. All participants will undergo a thorough assessment at baseline, and at 12 weeks post-baseline.

DETAILED DESCRIPTION:
Auditory hallucinations represent some of the most frequent and debilitating symptoms in schizophrenia spectrum disorders (SSD), affecting up to 80 % of individuals with SSD. Despite receiving treatment with antipsychotic medication, nearly one-third of these individuals continue to experience psychotic symptoms.

Virtual Reality-based interventions have emerged to address the essential need for targeted and effective psychotherapeutic interventions for auditory hallucinations. A recent randomized controlled trial (RCT) has developed and tested a fully immersive Virtual Reality-based intervention, with preliminary results indicating that this approach is effective in mitigating the severity of auditory hallucinations.

The Neuro-VR study aims to improve the effectiveness of this Virtual Reality-based intervention by incorporating real-time EEG-based neurofeedback into the intervention. We expect that augmenting the VR-based intervention with EEG-based neurofeedback will improve both its tolerability and effectiveness by using individual neurophysiological responses to guide the intervention.

The primary objective of the pilot study is to evaluate whether the combination of Virtual Reality and EEG-based neurofeedback is a feasible and acceptable therapeutic approach for treating auditory hallucinations in SSD. A secondary objective is to investigate whether Virtual Reality combined with EEG-based neurofeedback provides indications of being superior to Virtual Reality alone in reducing severity of auditory hallucinations, improving daily functioning and enhancing quality of life in individuals with SSD.

If the pilot study is found successful it could pave the way for broader clinical trials to document the effect of augmenting Virtual Reality-based interventions with real-time feedback from neurophysiological responses. In the long run, this combined approach can be implemented in the mental health clinics to complement traditional treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Age of 18-65 years
3. Diagnosis of schizophrenia spectrum disorder (ICD-10 codes: F20, F22-23; F25-29)
4. Symtoms of Auditory Verbal Hallucinations within at least the past 3 months (corresponding to SAPS score of 3 or more)
5. Identification of at least one dominant voice
6. No changes in antipsychotic medications four weeks prior to inclusion in the project
7. No planned changes in antipsychotic medication in the 12 weeks following inclusion in the project
8. A command of Danish or English sufficient to engage in therapy

Exclusion Criteria:

1. Rejecting informed consent
2. A diagnosis of organic brain disease
3. Intellectual disability (IQ ˂ 70)
4. A primary diagnosis of substance dependence hindering engaging in therapy
5. Hear voices in a language the therapist does not speak
6. Inability to tolerate the therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability as assessed by recruitment rate | Recruitment rate is monitored throughout the study period (1 year)
  Percentage of target sample (30 participants) recruited after 12 months from study start.
Feasibility and acceptability to the VR-NF intervention as assessed by retention rate | Retention rates are monitored throughout the study period (1 year)
  Percentage of included participants in the experimental group who retent to treatment at cessation of therapy (8 sessions).
Feasibility and acceptability to the VR-NF intervention as assessed by level of satisfaction in the experimental group | At 12 weeks follow up
  Percentage of participants in the experimental group reporting a satisfaction rating of more than 7 on a Likert scale ranging from 1-10 with higher scoring indicating a higher level of satisfaction with therapy.

SECONDARY OUTCOMES:
Severity of positive symptoms (hallucinations, delusions, bizarre behavior and positive formal thought disorder) as assessed by the Scale for the Assessment of Positive Symptoms (SAPS) | Baseline and at 12 weeks follow up
  SAPS is an interviewer-administered instrument with 34 items measuring positive symptoms in schizophrenia. Each item is rated on a 6-point scale ranging from None (0) to Severe (5) with higher scoring reflecting greater severity of positive symptoms.
Severity of auditory hallucinations as assessed by The Psychotic Symptom Rating Scales, Auditory Hallucination subscale (PSYRATS-AH) | Baseline and at 12 weeks follow up
  PSYRATS-AH is an interviewer-administered instrument with 11 items assessing characteristics of hallucinations: frequency; duration; location; loudness; beliefs about origin of voices; amount of negative content of voices; degree of negative content; amount of distress; intensity of distress; disruption and control.
  Each item is rated on a 5-point scale (0-4) with higher scores reflecting greater severity of auditory hallucinations.
  Additionally, an optional item measuring Number of Voices will be included.
Level of acceptance of and action in relation to the hallucinated voices as assessed by the Voices Acceptance and Action Scale (VAAS) | Baseline and at 12 weeks follow up
  The VAAS is a self-report scale assessing level of acceptance of and action in relation to the hallucinated voices rated on a 5-point Likert scale ranging from 'Strongly Disagree' (1) to 'Strongly Agree' (5) with higher scores reflecting higher levels of acceptance and action in relation to the hallucinated voices.
Beliefs about voice power, voice intent and responding styles as assessed by the revised Beliefs about Voices Questionnaire (BAVQ-R) | Baseline and at 12 weeks follow up
  The BAVQ-R is a self-report questionnaire assessing beliefs about hallucinated voices. Each item is rated on a 4-point scale ranging from Disagree (0), Unsure (1), Slightly agree (2), Strongly agree (3) with higher scores indicating greater endorsement of a belief.
Level of perceived power in relation to the hallucinated voice as assessed by the Voice Power Differential Scale (VPDS) | Baseline, 1 week post baseline, 8 weeks post baseline and at 12 weeks follow up
  The VPDS is a self-report questionnaire with seven items rated on a 5-point scale (1-5) with a total score ranging from 7-35. Higher scores indicate that the voice is perceived to have greater power compared to the respondent.
  At therapy sessions 1 and 8, the participants will be asked to complete the questionnaire focusing on the hallucinated voice they choose to focus on during therapy.
Responding styles to hallucinated voices as assessed by the Assertive Responding to Voices (Approve - Voices) questionnaire | Baseline, 1 week post baseline, 8 weeks post baseline and at 12 weeks follow up
  The Assertive Responding to Voices (Approve - Voices) questionnaire comprises 15 items assessing different ways to respond to the hallucinated voices.
  Scores range from 0-10 with higher scores indicating higher degree of the specific responding to voices.
  At therapy sessions 1 and 8, the participants will be asked to complete the questionnaire focusing on the hallucinated voice they choose to focus on during therapy.
Social and daily functioning as assessed by the Personal and Social Performance Scale (PSP) | Baseline and at 12 weeks follow up
  The PSP is an interviewer administered instrument assessing different domains of social and daily functioning: job/education, social relations, personal hygiene and aggressive behaviour.
  A total score ranges from 1-100 with higher scores indicating a higher degree of functioning.
Social functioning as assessed by the Social Functioning Scale (SFS) | Baseline and at 12 weeks follow up
  The SFS is a self-report instrument assessing social functioning among individuals with schizophrenia.
  The instrument comprises seven domains: Social engagement/withdrawal, Interpersonal behaviour, Prosocial activities, Recreation, Independence-competence, Independence-performance and Employment/occupation.
  The minimum raw score is 0 and maximum raw score is 223 with higher scoring indicating a higher level of functioning.

OTHER OUTCOMES:
Level of negative symptoms as assessed by the Brief Negative Symptoms Scale (BNSS) | Baseline and at 12 weeks follow up
  The BNSS is a an interviewer-administered instrument comprising 13 items and five domains of negative symptoms: anhedonia, asociality, avolition, blunted effect and alogia.
  Each item is rated on a 7-point scale (0-6) with higher scores reflecting a higher level of negative symptoms.
Level of negative symptoms as assessed by the Self Evaluation of Negative Symptoms (SNS) | Baseline and at 12 weeks follow up
  The SNS is a self-report questionnaire with 20 items rated on 3-point scale ranging from Strongly agree (2) to Strongly disagree (0). A total score ranges from 0 to 40 with higher scoring reflecting a higher degree of self-evaluated negative symptoms.
Ability to use emotion regulation strategies as assessed by the Emotion Regulation Questionnaire (ERQ) | Baseline and at 12 weeks follow up
  The ERQ is a self-report questionnaire with 10 items that measure the extent to which the respondent regulates and manages emotions using two different strategies: cognitive reappraisal and expressive suppression.
  Each item is rated on a 7-point scale ranging from Completely disagree (1) to Completely agree (7).
  The two subscales are scored separately with higher scores reflecting greater use of the specific strategy.
Difficulties in emotion regulation as assessed by the Difficulties in Emotion Regulation Scale, short version (DERS-16) | Baseline and at 12 weeks follow up
  The DERS-16 is a self-report questionnaire with 16 items assessing different dimensions of emotion regulation difficulties: Nonacceptance of negative emotions, Inability to engage in goal-directed behaviors when distressed, Difficulties controlling impulsive behaviors when distressed, Limited access to emotion regulation strategies perceived as effective and Lack of emotional clarity.
  Each item is rated on a 5-point Likert-scale ranging from Almost never (1) to Almost always (5). A total score is calculated by summing the scores of the different subscales ranging from 16 to 80 with higher scores reflecting greater levels of emotion dysregulation.
Beliefs about self and others as assessed by The Brief Core Schema Scales: Beliefs about self and others (BCSS) | Baseline and at 12 weeks follow up
  The BCSS is a self-report questionnaire with 24 items assessing four dimensions of schemata concerning self and others: Negative-self, Positive-self, Negative-others and Positive-others.
  Each item is rated on a 5-point scale ranging from No (0) to Believe it totally (4) with higher scores indicating greater endorsement of a schema.
Level of client satisfaction with intervention as assessed by the Client Satisfaction Questionnaire (CSQ) | At 12 weeks follow up
  The CSQ is a self-report questionnaire with 8 items measuring client satisfaction with the intervention.
  Each item is scored on a 4-point scale ranging from 1-4 with higher scores reflecting greater satisfaction with intervention.
Level of simulator sickness elicited by virtual reality as assessed by the Simulator Sickness Questionnaire (SSQ) | 2, 4 and 8 weeks post baseline
  The SSQ is a self-report questionnaire with 16 items measuring different symptoms of simulator sickness. Each item is rated on a 4-point scale ranging from None (0) to Severe (3) with higher scores indicating a higher level of symptoms.
Level of depressive symptoms as assessed by the Calgary Depression Scale for Schizophrenia (CDSS) | Baseline and at 12 weeks follow up
  The CDSS is an interviewer-administered instrument comprising 9 items assessing level of depression among individuals with schizophrenia. Each item is rated on a 4-point scale ranging from Absent (0) to Severe (3) with higher scores indicating a higher level of depressive symptoms.
Severity of suicidal ideation and risk for suicidal behavior as assessed by the Suicidal Ideation Attributes Scale (SIDAS) | Baseline and at 12 weeks follow up
  The SIDAS is a self-report questionnaire with 5 items measuring different aspects of suicidal thoughts: frequency, controllability, closeness to attempt, level of distress associated with the thoughts and impact on daily functioning.
  Each item is rated on a 11-point scale ranging from 0-10 with higher scores reflecting greater severity of suicidal thoughts.
Experience with childhood traumas as assessed by the Childhood Trauma Questionnaire(CTQ) | Baseline
  The CTQ is a retrospective, self-report questionnaire with 28 items measuring traumatic experiences in childhood.
  Each item is rated on a 5-point Likert scale ranging from Never (1) to Very often (5) with higher scores reflecting greater severity of childhood trauma.
Psychological well-being as assessed by The World Health Organisation- Five Well-Being Index (WHO-5) | Baseline and at 12 weeks follow up
  The WHO-5 is a self-report questionnaire with 5 items measuring subjective psychological well-being. Each item is scored on a 6-point scale ranging At no time (0) to All of the time (5).
  A total raw score is ranging from 0 to 25. To calculate the final score, the total raw score is multiplied by 4 with higher scores reflecting higher levels of well-being.
Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline and at 12 weeks follow up
  The PSQI is a self-report questionnaire measuring sleep quality and disturbances over a 1-month time.
  The questionnaire consists of a combination of Likert- type and open-ended questions with higher scores indicating higher level of sleep disturbances.
Level of self-efficacy as assessed by the General Self-Efficacy Scale (GSE) | Baseline and at 12 weeks follow up
  The GSE is a self-report questionnaire with 10 items meausering percevied self-efficacy. Each item is rated on a 4-point scale ranging from Not at all true (1) to Exactly true (4) with higher scores reflecting greater self-efficacy.
  Total score ranges from 10 to 40.
Level of insight into illness as assessed by the Birchwood Insight Scale (BIS) | Baseline and at 12 weeks follow up
  The BIS is a self-report questionnaire with 8 items measuring insight in mental illness. Each item is rated on a 3-point scale ranging from Agree, Disagree to Unsure.
  A total score is calculated by summing the scores of three subscales (Awareness of symptoms, Awareness of illness and Need for treatment) and ranges from 0-12 with higher scores reflecting greater insight into illness.
Readiness for therapy as assessed by the Readiness for Therapy Questionnaire (RTQ) | Baseline
  The RTQ is a self-report questionnaire with 6 items measuring positive attitude and preparedness to enter therapy.
  Each item is rated on a 5-point Likert scale ranging from Strongly disagree (0) to Strongly agree (4).
  Items 2, 3 and 6 are reversed scored. A higher score reflects greater readiness for therapy.
Change in EEG (Electroencephalography) activity - P50 suppression | Baseline and at 12 weeks follow up
  P50 suppression is a measure of sensory gating that can be assessed by measuring electroencephalographic (EEG) responses to repeated pairs of auditory clicks The participants will be instructed to count auditory clicks, either in pairs or individually, while keeping the eyes closed.
  The paradigm will last for a total of 21 minutes, divided into 3 intervals of 7 minutes each.
Change in EEG (Electroencephalography) activity - Mismatch Negativity (MMN) | Baseline and at 12 weeks follow up
  The mismatch negativity (MMN) is a brain response to violations of a rule, established by a sequence of sensory stimuli. The participants will watch a movie on a screen while hearing some pure tones. The participants will be instructed to try to ignore the tones and not react on them, sitting as still as possible.
  This paradigm lasts 12 minutes.
Change in EEG (Electroencephalography) activity - Auditory Steady State Response (ASSR) | Baseline and at 12 weeks follow up
  ASSRs are evoked brain responses to repeated auditory stimulus. A sequence of tones is repeatedly presented to the participants. The participants are instructed to keep their gaze fixed on a cross displayed on a screen in front of them while they sit as still as possible.
  This paradigm lasts 6 minutes.
Change in EEG (Electroencephalography) activity - Selective Attention (SA) | Baseline and at 12 weeks follow up
  A Selective Attention (SA) paradigm will measure the ability to focus on relevant information, while filtering out distracting information.
  The participants will be presented to standard auditory stimuli, followed by a deviant stimulus with a higher frequency across both ears. The participants will be instructed to press a button if they hear a deviant stimulus on a specific ear.
Change in EEG (Electroencephalography) activity - Resting State | Baseline and at 12 weeks follow up
  EEG recordings at resting state will measure spontaneous neural activity. The participants will be instructed to sit as still as possible while keeping their eyes open and fixed on a cross displayed on a screen in front of them. The participants will be instructed to not think of anything in specific.
  This paradigm will last 5 minutes.
A qualitative measure of feasibility and acceptability to the VR-NF intervention | Semi-structured interviews will be conducted throughout the study period (up to 18 months)
  Qualitative semi-structured interviews with participants and therapists will be conducted to investigate their experiences with the experimental intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Louise B. Glenthøj, DMSc, PhD, Principal Investigator — Copenhagen Research Center for Mental Health - CORE
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Copenhagen, Hellerup, Denmark